CLINICAL TRIAL: NCT03411772
Title: Impact of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Pain After Laparoscopic Bariatric Surgery: a Randomized Double Blind Controlled Trail
Brief Title: Trial on TAP Block After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mansourau44
Record Dates: First submitted 2018-01-14; First posted 2018-01-26 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients will sign an informed consent entailing their knowledge and acceptance of being included in the trial, however patients will not be aware to the group they will be included to. In addition, the operating surgeon will not be aware to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): Patients undergoing bariatric surgery having TAP block upon completion of the procedure
  Interventions: Procedure: TAP block; Procedure: Bariatric surgery
- Non TAP block (Sham Comparator): Patients undergoing bariatric surgery without having TAP block
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: TAP block — Injection of 20 mL of 0.25% bupivacaine in the transversus abdominis plane under ultrasound guidance after performing bariatric surgery
  Arms: TAP block
Procedure: Bariatric surgery — Bariatric surgery will be conducted

SUMMARY:
Patients undergoing bariatric surgery will be divided randomly into two groups: the first will have TAP block upon completion of surgery and the second groups will not have TAP block.

DETAILED DESCRIPTION:
Upon completion of the laparoscopic bariatric procedure to be performed for every patient and just before recovery from general anesthesia, an ultrasound-guided TAP block will be conducted in the operative theater by the anesthetist for group I patients whereas group II will be recovered from anesthesia without having a TAP block.

The ultrasound probe will be placed on the lateral abdominal wall in the mid-axillary line between the lower costal margin and iliac crest. Using ultrasound will allow accurate deposition of the local anesthetic in the correct neurovascular plane. A spinal needle will be advanced using in-plane technique between the aponeurosis of the internal oblique and transversus abdominis muscles. With intermittent aspiration, 20 mL of local anesthetic (0.25% bupivacaine) will be deposited in the TAP on each side and seen as a hypoechoic shadow pushing the two layers apart.

ELIGIBILITY:
Inclusion Criteria:

* All morbidly obese patients of both genders with BMI >35 kg/m2 who will be admitted to the General Surgery Department within the study period to undergo laparoscopic bariatric procedures will be included in this study. Bariatric procedures to be performed will comprise LSG, roux en-Y- gastric bypass, mini-gastric bypass, gastric plication, and single anastomosis sleeve ileal (SASI) bypass.

Exclusion Criteria:

* Patients unfit for general anesthesia, patients with secondary obesity due to endocrine disorders, patients with psychiatric disorders, patients with drug abuse or history of opioid intake or chronic pain disorder, patients with contraindication to peripheral nerve block such as allergy to local anesthetics and coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative abdominal pain | first 24 hours after surgery
  Degree of postoperative pain measured by Visual Analogue Scale from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No